CLINICAL TRIAL: NCT06579963
Title: A Randomized Controlled Trial (RCT) Evaluating the Effects of Cool Roofs on Health Outcomes Using Smartwatches: a Global Multi-center Study
Brief Title: Assessing the Effect of Cool Roofs on Health Using Smartwatches
Acronym: REFLECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aditi Bunker (Other)
Collaborators: Sika Services AG (Unknown); SOPREMA (Unknown); Engineered Polymer Solutions (EPS B.V.) (Unknown); Resene (Industry); Pacific Community (Other); Habitat for Humanity (Other); The Tindall Foundation (Other); Labfront (Industry); Instituto Tecnológico de Hermosillo (Unknown); University of Ouagadougou, Burkina Faso (Other); Indian Institute of Public Health, India (Other); Boston University (Other); Rutgers University (Other); London School of Hygiene and Tropical Medicine (Other); Heidelberg University (Other)
Responsible Party: Sponsor-Investigator, Aditi Bunker, Co-Principal Investigator, University of Auckland, New Zealand
Organization: University of Auckland, New Zealand (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3728163; 226745/Z/22/Z (Other Grant/Funding Number: Wellcome Trust UK)
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Heart Rate; All-day Steps; Distance Walked; Active Minutes; Moderate-intensity Activity Minutes; Vigorous-intensity Activity Duration; Sleep Quantity; Time in Sleep Stages; Awake Duration; Sleep Score
Keywords: Hot Temperature; Humidity; Housing; Wearable; Smartwatch; Heart rate; Cardiovascular; Physical activity; Sleep; Cool roof; Heat stress
MeSH Terms: conditions — Motor Activity; Heat Stress Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Trial participants will be aware of the intervention to which they have been allocated, and the research fieldworkers will be aware of the intervention allocation. The trial steering committee members and trial statistician will remain blinded until the end of trial period and data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cool roof (Experimental): Households will receive sunlight reflecting 'cool roof' coating on their roofs.
  Interventions: Other: Cool roof
- No cool roof (No Intervention): No cool roof application. Households will keep their original roofing for the duration of the trial.

INTERVENTIONS:
Other: Cool roof — Cool roofs are a sunlight reflecting roof coating that can reduce indoor temperature. Cool roofs have high solar reflectance (reflecting the ultraviolet and visible wavelengths of sunlight, reducing heat transfer to the surface of a roof) and high thermal emittance (radiating absorbed solar energy).
  Arms: Cool roof

SUMMARY:
Ambient air temperatures in Asian, Latin American, African, and Pacific climate hotspots have broken record highs in 2024. Solutions are needed to build heat resilience in communities and adapt to increasing heat from climate change. Sunlight-reflecting cool roof coatings may passively reduce indoor temperatures and energy use to protect home occupants from extreme heat. Occupants living in poor housing conditions globally - for example in informal settlements, slums, and low-socioeconomic households - are susceptible to increased heat exposure.

Heat exposure can instigate and worsen numerous physical, mental and social health conditions. The worst adverse health effects are experienced in communities that are least able to adapt to heat exposure. By reducing indoor temperatures, cool roof application may improve heart health, sleep and physical activity in household occupants.

The long-term research goal is to identify viable passive housing adaptation technologies with proven health benefits to reduce the burden of heat stress in communities affected by heat globally. To meet this goal, the investigators will use smartwatches to measure the effects cool roof application on heart health, sleep and physical activity in four urban climate hotspots: Ouagadougou, Burkina Faso; Hermosillo, Mexico; Ahmedabad, India; and Niue, Oceania.

DETAILED DESCRIPTION:
Increasing heat exposure from climate change is causing and exacerbating heat-related illnesses in millions worldwide - particularly in low resource settings. June 2024 was the 13th consecutive hottest month on record globally - shattering previous records. Heat exposure can instigate and worsen numerous health conditions. Adaptation is essential for protecting people from increasing heat exposure. The built environment, especially homes, are ideal for deploying interventions to reduce heat exposure and accelerate adaptation efforts. However, evidence is currently lacking on a global scale - generated through empirical studies - guiding the uptake of interventions to reduce indoor heat stress in low resource settings.

Sunlight-reflecting cool roof coatings passively reduce indoor temperatures and lower energy use, offering protection to home occupants from extreme heat. Continuous monitoring of health and wellbeing using smartwatches can provide insight into important parameters such as heart rate, sleep and physical activity - which are all affected by heat. Using smartwatches, the investigators will also continuously measure health and wellbeing outcomes during the day and night. The investigators will conduct a global multi-centre study to investigate the effects of cool-roof use on heart rate, sleep and physical activity in four urban climate hotspots - Ouagadougou, Burkina Faso (sub-Saharan Africa), Ahmedabad, India (Asia), Niue (Oceania), and Sonora, Mexico (Latin America). These sites represent hotspots where people experience a triple burden from heat exposure, chronic health issues and vulnerable housing conditions (slums, informal settlements and low socioeconomic housing). They also exhibit diversity in climate profiles, housing typology, level of socioeconomic development, population density and rates of urbanisation.

This trial will quantify whether cool roofs are an effective passive home cooling intervention with beneficial health effects for vulnerable populations in four locations. Findings will inform global policy responses on scaling cool roof implementation to protect people from increasing heat exposure driven by climate change.

ELIGIBILITY:
Inclusion Criteria:

* Permanent household resident

Exclusion Criteria:

* Roof damage, inaccessible or instability of roof adversely affecting cool roof coating application.
* Participant unable to provide written/verbal informed consent. Participants will be excluded if they are not willing or able to wear a smartwatch.
* In Mexico and Niue, participants will be excluded if they do not have a smartphone with an internet connection that can connect to the smartwatch.
* Only one participant per household.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Heart rate in beats per minute measured at 15-second intervals using Garmin Vivosmart 5 devices.

SECONDARY OUTCOMES:
All-day steps | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The number of steps measured daily using Garmin Vivosmart 5 devices.
Active minutes | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The total number of minutes of active exercise daily using Garmin Vivosmart 5 devices.
Distance walked | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The total distance walked daily using Garmin Vivosmart 5 devices.
Moderate-intensity activity minutes | MeasuSmartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at barements will be taken continuously for 12 months. Participants will be asked to wear their smartwatch for at least two weeks every month.
  The total number of minutes of moderate-intensity activity daily using Garmin Vivosmart 5 devices.
Vigorous-intensity activity duration | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The total number of minutes of vigorous-intensity activity daily using Garmin Vivosmart 5 devices.
Sleep quantity | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The number of hours spent asleep each night using Garmin Vivosmart 5 devices.
Time in sleep stages | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The number of hours spent in sleep stages each night using Garmin Vivosmart 5 devices.
Awake duration | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The number of hours spent awake during sleep time each night using Garmin Vivosmart 5 devices.
Sleep score | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The Garmin sleep score (0-100) each night using Garmin Vivosmart 5 devices. A higher score means a better outcome.

CONTACTS AND LOCATIONS:
Locations (4):
- University Joseph Ki-Zerbo, Ouagadougou, Burkina Faso
- Indian Institute of Public Health Gandhinagar, Ahmedabad, Gandhinagar, India
- Instituto Tecnológico de Hermosillo, Hermosillo, Sanora, Mexico
- Niue, Alofi, Niue

IPD SHARING:
Plan to Share IPD: Yes
Data that can be shared unconditionally underpinning the published research articles will be made available to other researchers at the time of publication, and data will be linked via the article DOI. Data that cannot be unconditionally shared upon publication owing to confidentiality or data protection requirements will be identified as such and a contact email will be provided in relevant publications for data access enquiries by other researchers. Individual names of study participants and identifying factors will be removed prior to data sharing.
  It is expected that demographic data of people at the study sites (family size and composition, basic socioeconomic indicators) may contain personally identifiable information and location data. All such data will be removed prior to storage on online data repositories and therefore will be available to be publicly shared at the time of publication of manuscripts.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the time of publication.
URL: http://reflect.org.nz